CLINICAL TRIAL: NCT04160819
Title: The Effects of Individualized Nutritional Intervention Program in Malnutrition Elderly With Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pei-Hsin Yang (Other)
Responsible Party: Sponsor-Investigator, Pei-Hsin Yang, investigator, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201700126B0C501
Record Dates: First submitted 2019-11-07; First posted 2019-11-13 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Pneumonia
Keywords: nutritional intervention; malnutrition; respiratory disease
MeSH Terms: conditions — Pneumonia; Malnutrition; Respiration Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individualized nutritional intervention programs (iNIPs) (Experimental): Participants in the NI group received an iNIP according to energy and protein intake requirements in addition to dietary advice based on face-to-face interviews with their family members during hospitalization. After discharge, phone calls are adopted for prescribing iNIPs. Anthropometry (i.e., body mass index, limb circumference, and subcutaneous fat thickness), blood parameters (i.e., albumin and total lymphocyte count), hospital stay, Mini-Nutritional Assessment-Short Form (MNA-SF) score, target daily calorie intake, total calorie intake adherence rate, and three-major-nutrient intake were assessed during hospitalization and 3 and 6 months after discharge. Both groups received regular follow-up through phone calls. Furthermore, the rate of readmission resulting from pneumonia was recorded after discharge.
  Interventions: Other: Assigned Interventions
- standard care (SC) group (No Intervention): SC group was only provided standard nutritional supplements according to the Kaohsiung Chang Gung Memorial Hospital Nutrition Department, and patients' family members were not provided dietary advice.

INTERVENTIONS:
Other: Assigned Interventions — Participants in the NI group received an iNIP according to energy and protein intake requirements in addition to dietary advice based on face-to-face interviews with their family members during hospitalization. After discharge, phone calls are adopted for prescribing iNIPs.
  Other Names: The SC group was only provided standard nutritional supplements , and patients' family members were not provided dietary advice.
  Arms: individualized nutritional intervention programs (iNIPs)

SUMMARY:
To investigate the effects of an individualized nutritional intervention programs (iNIPs) on nutritional status and readmission rate in older adults with pneumonia during hospitalization and 3 and 6 months after discharge.

DETAILED DESCRIPTION:
Method: Eighty-two malnourished older adults with primary diagnosis of pneumonia participated. Patients were randomly allocated to either a nutrition intervention (NI) group or a standard care (SC) group. Participants in the NI group received an iNIP according to energy and protein intake requirements in addition to dietary advice based on face-to-face interviews with their family members during hospitalization. After discharge, phone calls are adopted for prescribing iNIPs. Anthropometry (i.e., body mass index, limb circumference, and subcutaneous fat thickness), blood parameters (i.e., albumin and total lymphocyte count), hospital stay, Mini-Nutritional Assessment-Short Form (MNA-SF) score, target daily calorie intake, total calorie intake adherence rate, and three-major-nutrient intake were assessed during hospitalization and 3 and 6 months after discharge. Both groups received regular follow-up through phone calls. Furthermore, the rate of readmission resulting from pneumonia was recorded after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of pneumonia by a physician
* Age more than 65 years
* Malnutrition status indicated by body mass index (BMI) <18.5 kg/m2 or Mini-Nutritional Assessment-Short Form (MNA-SF) score≤7

Exclusion Criteria:

* Renal insufficiency (glomerular filtration rate [GFR] <60 mL/min/1.73 m2 or GFR staging of G3b-G5)
* Cancer
* Hospital stay <7 days

Ages: 66 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
nutritional status | up to 6 months of intervention
  Mini-Nutritional Assessment short-form scores;MNA-SF scores ranging within 0-7, 8-11, and 12-14 indicate malnutrition, risk of malnutrition, and normal nutritional status, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Pei-Hsin Yang, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Currently in the submission stage, and then share with other researchers after publication.